CLINICAL TRIAL: NCT05329064
Title: A Single Arm Phase-IV Study to Determine Reactogenicity and Immunogenicity of Delayed COVID-19 Vaccine Schedule in Children
Brief Title: Determining Reactogenicity and Immunogenicity of Delayed COVID-19 Vaccine Schedule in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/2003
Record Dates: First submitted 2022-04-11; First posted 2022-04-14 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-03

CONDITIONS: Vaccine Reaction; COVID-19; Children, Only
Keywords: COVID-19; Vaccine; Children
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10mcg of BNT162b2 (Pfizer-BioNTech/Comirnaty®) (Other): 10mcg of BNT162b2 (Pfizer-BioNTech/Comirnaty®) for each dose. Two doses will be given at 2 months apart between doses.
  Interventions: Biological: BNT162b2 Pfizer-BioNTech/Comirnaty

INTERVENTIONS:
Biological: BNT162b2 Pfizer-BioNTech/Comirnaty — The study will use 10mcg of BNT162b2 (Pfizer-BioNTech/Comirnaty®) for each dose.
  Two doses will be given at 2 months apart between doses.

SUMMARY:
COVID-19 vaccine response data in children 5 to 11 years old remain scarce. Our understanding of the safety and immune responses including humoral and cellular responses generated in children remains limited.

Safety of the vaccine is critical in the risk benefit assessment of vaccination in young children. Available data show a trend for increased risk of myocarditis after second dose, especially in males and younger age groups. It is unknown if reduced antigen dose will alter this risk in 5y to <12y age group. Reassuringly, data from early roll-out in the USA have not reported any safety signals to date. Alternate (reduce dosing or delayed dosing) strategies could help ensure maximum protection with reduced risk of side-effects. There is currently no data available to inform how long protection would last in the reduced dose or delayed dosing strategy.

The trial will inform the potential use of alternate dosing schedules such as single dose or delayed dose to minimise risk and maximise benefit of COVID-19 vaccination in children 5 to 11 years old.

DETAILED DESCRIPTION:
BNT162b2 (Pfizer-BioNTech/Comirnaty®) vaccine is a mRNA vaccine that is (26/11/2021) approved for use in adults and adolescents (12 years old and above) under the Pandemic Special Access Route (PSAR) by the Health Sciences Authority (HSA), Singapore.1 Two doses of vaccine (30mcg) given 3 weeks apart was shown to be > 95% effective in the prevention of symptomatic COVID-19 infection.2 The latest phase 3 trial of the vaccine using a lower (10 mcg) two dose schedule (3 weeks apart) in children aged 5 to 11 year old was found to be > 90% effective.

Older age groups and those with comorbidities such as obesity, diabetes mellitus, etc are at highest risk of severe COVID-19 disease. Currently, recommendations for vaccination have been extended to adolescents in Singapore as well as many countries including the USA, Israel and Ireland, in view of the high rates of infection in this age group. On 29 October 2021, the FDA authorised the use of BNT162b2 Pfizer-BioNTech/Cominarty vaccine for emergency use in children 5 to 11 years old.4 Subsequently, the CDC recommended COVID-19 vaccination of children 5 to 11 years old in the USA using intramuscular 10mcg of BNT162b2 Pfizer-BioNTech/Comirnaty®) vaccine given 3 weeks apart.

A key concern regarding paediatric vaccination is a rare side effect of inflammation of the heart muscle (myocarditis) that has been observed after receipt of the second dose of BNT162b2,especially in younger age groups including adolescents and males. Centre for Disease Control (CDC), USA reported that there were 9.8 cases of myocarditis per million first doses given and this rose to 67 per million after the second dose. Most cases of myocarditis were benign and self-limiting but long-term impact remains uncertain.

There are possible alternatives to a standard two dose schedule given 21 days apart which may help reduce the risk of adverse events such as myocarditis. The extended interval between doses had been shown in the UK to result in improved immunogenicity in adults. The optimum timing of such a delayed dosing schedule remains unknown in children and identifying the best timing to help delay the need for boosters in children will be useful.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 5 to 11 years old
* No contraindications to mRNA COVID-19 Pfizer-BioNTech vaccines
* Had never received any COVID-19 vaccine before
* Never had previous COVID-19 infections

Exclusion Criteria:

* Children outside the age group.
* Immunocompromised children.
* Participants with previous history of COVID-19 infection.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage neutralizing antibody levels at 2m | 2 Months
WHO International units/ml neutralizing antibody levels at 2m | 2 Months
Geometric mean titres (GMT) neutralizing antibody levels at 2m | 2 Months

SECONDARY OUTCOMES:
Percentage neutralizing antibody levels at 6m and 9 to 12m | 12 Months
WHO International units/ml neutralizing antibody levels at 6m and 9 to 12m | 12 Months
GMT neutralizing antibody levels at 6m and 9 to 12m | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Bukit Timah, Singapore

IPD SHARING:
Plan to Share IPD: Undecided